CLINICAL TRIAL: NCT03856203
Title: Longitudinal Assessment of Nutrition Status of Adults With PKU Before and During Treatment With Pegvaliase
Brief Title: Nutrition Status of Adults With PKU Before and During Treatment With Pegvaliase
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Krista Viau, Principal Investigator, Boston Children's Hospital
Other Study IDs: IRB-P00029889
Record Dates: First submitted 2019-02-14; First posted 2019-02-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Conduct a prospective, longitudinal study to evaluate nutritional status in adults with phenylketonuria (PKU) before and during treatment with pegvaliase (Palynziq™).

DETAILED DESCRIPTION:
The investigators will compare intra-subject change in adults with PKU who follow a protein-restricted diet (protein intake less than the RDA for protein based on weight (0.8 g/kg/day) with or without a PKU medical food) within 90 days of starting pegvaliase (baseline) and 9 and 15 months later. The investigators will collect laboratory measures of nutrition status, anthropometrics, Dual-Energy X-Ray Absorptiometry (DXA) to measure body composition and bone mineral density (BMD), and indirect calorimetry to measure resting energy expenditure (REE). In addition, three-day food records will be obtained to assess protein intake and overall diet quality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of phenylketonuria
* Aged 18-65 years
* Following a protein-restricted diet with or without medical food within the last 30 days
* Routine natural protein intake from food is less than the RDA for protein based on weight (0.8 g/kg/day).
* If not consuming animal proteins, recommended protein intake is 115% RDA due to lower bioavailability of plant proteins.
* Within ±90 days of starting treatment with pegvaliase at time of study enrollment

Exclusion Criteria:

* Unable to consent to study
* Under age 18 or over age 65 years
* Routine natural protein intake is greater than the RDA for protein (0.8 g/kg/d) within the last 30 days.
* Females who are currently pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit adults with PKU who are starting therapy with pegvaliase and currently following a protein-restricted diet with or without medical food.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Intra-subject change in intact and medical food protein intake (grams/day) as reported on three-day food records at months 0, 9, and 15. | 15 months
Intra-subject change in serum markers of protein status at months 0, 9, and 15. | 15 months
Intra-subject difference in lean body mass (%LBM) from month 0 to 15. | 15 months
Intra-subject difference in bone mineral density from month 0 to 15. | 15 months

SECONDARY OUTCOMES:
Intra-subject change in concentrations of serum markers of micronutrient status at months 0, 9, and 15. | 15 months
Intra-subject change in serum concentrations of essential fatty acid nutriture at months 0, 9, and 15. | 15 months
Intra-subject change in BMI at months 0, 9, and 15. | 15 months
Intra-subject change in serum markers of cardiovascular status at months 0, 9, and 15. | 15 months
Intra-subject change in emotional eating, cognitive restraint, uncontrolled eating at months 0, 9, and 15. | 15 months
  Three-Factor Eating Questionnaire (TFEQ)-18 is an 18-item questionnaire measured on a four-point scale cognitive restraint (6 items), uncontrolled eating (9 items) and emotional eating (3 items). Responses are measured on a four-point scale and the raw scores for each subscale are transformed to correspond to a 0-100 point scale. Higher scores in the respective scales are indicative of greater cognitive restraint, emotional eating, and uncontrolled eating.
Intra-subject change in food neophobia at months 0, 9, and 15. | 15 months
  Food Neophobia Scale, which was adapted for a PKU population, includes nine questions measured on a seven-point scale with a higher total score indicative of greater food neophobia (score range 9-63).
Intra-subject change in Epicurean eating tendencies at months 0, 9, and 15. | 15 months
  Epicurean eating tendencies questionnaire includes seven items measured with a seven-point scale (range 7-49). Higher scores indicative of greater Epicurean eating tendencies.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No